CLINICAL TRIAL: NCT03165097
Title: A Single-center, Double-blind, Parallel-group, Randomized, Placebo-controlled, Multiple-ascending Oral Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT-709478 in Healthy Subjects
Brief Title: Study to Evaluate Safety and Tolerability of ACT-709478 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AC-083-102; 2017-000336-34 (EudraCT Number)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Healthy Subjects
Keywords: tolerability; safety
MeSH Terms: interventions — ACT-709478; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ACT-709478 (Experimental): 40 subjects will receive multiple doses of ACT-709478 at the planned dose levels of 30, 60, 100, and 200 mg.
  Each dose level will be investigated in a new cohort of 10 healthy male and female subjects (4 male subjects on active drug and 1 on placebo, 4 female subjects on active drug and 1 on placebo) undergoing one treatment period with a once daily dosing scheme.
  Interventions: Drug: ACT-709478
- Placebo (Placebo Comparator): Matched placebo administered accordingly
  Interventions: Drug: Placebo
- Midazolam (Other): 4 mg taken by mouth on Day 1 of the corresponding cohort
  Interventions: Drug: Midazolam
- ACT-709478 combined with Midazolam (Experimental): On Day 22 and Day 30, midazolam (4 mg) and ACT-709478 (60 mg or 100 mg) to be co-administered.
  Interventions: Drug: ACT-709478 combined with midazolam

INTERVENTIONS:
Drug: ACT-709478 — Hard gelatine capsules for oral administration
  Arms: ACT-709478
Drug: Placebo — Placebo capsules matching ACT-709478 capsules
  Arms: Placebo
Drug: Midazolam — Midazolam oral solution (2 mg/mL) applied with a syringe
  Arms: Midazolam
Drug: ACT-709478 combined with midazolam — Hard gelatine capsules for oral administration (ACT-709478) to be taken first followed by Midazolam oral solution (2 mg/mL) applied with a syringe
  Arms: ACT-709478 combined with Midazolam

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of ascending multiple doses of ACT-709478 in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Healthy male and female subjects aged between 18 and 55 years (inclusive) at screening
* Negative serum pregnancy tests at screening and negative urine pregnancy test at Day -1 for women and agreement to use 2 reliable methods of contraception for at least 3 months after last study drug administration
* Body mass index of 18.0 to 29.9 kg/m2 (inclusive) at screening
* Systolic blood pressure 100-140 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 50-90 bpm (inclusive), measured after 5 minutes in the supine position at screening and on Day -1
* Healthy on the basis of physical examination, cardiovascular, ophthalmological, neurological assessments and laboratory tests

Exclusion Criteria:

* Known hypersensitivity to ACT-709478 or drugs of the same class, or any of their excipients
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism, or excretion of the study treatments
* QT interval corrected with Fridericia's formula (QTcF) > 450 ms (using the ECG machine HR correction method) at screening and on Day -1
* Treatment with another investigational treatment within 2 months or 5 t1/2 (whichever is the longest) prior to screening or participation in more than four investigational treatment studies within 1 year prior to screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to Day 23
  The percentage of subjects with treatment-emergent adverse events will be reported
Changes from baseline in vital signs | up to Day 23
  Vital signs include diastolic and systolic blood pressure and pulse rate
Incidence of any clinical relevant findings in ECG variables | up to Day 23
  The number of subjects with any treatment-emergent electrocardiogram (ECG) abnormalities will be reported

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-709478 | up to Day 23
  Cmax is derived from the observed plasma concentration-time curves
Time to reach Cmax (tmax) of ACT-709478 | up to Day 23
  tmax is directly derived from the observed plasma concentrations
Terminal half-life (t1/2) of ACT-709478 | up to Day 23
  t1/2 is calculated from the terminal rate constant obtained from the plasma concentrations-time curves
Area under the plasma concentration-time curve AUC(tau) of ACT-709478 | up to Day 23
  AUCtau is defined as the area under the plasma concentration-time curve during one dosing interval
Area under the plasma concentration-time curve AUC(tau) of midazolam | 24 hours after dosing on Day 1, Day 22 and Day 30
  AUCtau is defined as the area under the plasma concentration-time curve during one dosing interval
Time to reach Cmax (tmax) | 24 hours after dosing on Day 1, Day 22 and Day 30
  tmax is directly derived from the observed plasma concentrations
Maximum plasma concentration (Cmax) of ACT-709478 | 24 hours after dosing on Day 1, Day 22 and Day 30
  Cmax is derived from the observed plasma concentration-time curves

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Parexel, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richard M, Kaufmann P, Ort M, Kornberger R, Dingemanse J. Multiple-Ascending Dose Study in Healthy Subjects to Assess the Pharmacokinetics, Tolerability, and CYP3A4 Interaction Potential of the T-Type Calcium Channel Blocker ACT-709478, A Potential New Antiepileptic Drug. CNS Drugs. 2020 Mar;34(3):311-323. doi: 10.1007/s40263-019-00697-1. PMID 31994022